CLINICAL TRIAL: NCT05076981
Title: Progesterone Levels During Ovulation and Luteal Phase in Spontaneous Natural Ovulatory Cycles vs Modified Natural Cycle. A Prospective Study
Brief Title: Progesterone Levels During Ovulation and Luteal Phase
Status: Completed | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Laura Melado, Principal Investigator, ART Fertility Clinics LLC
Other Study IDs: 2107-ABU-009-LM
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Infertility, Female
Keywords: luteal phase; natural cycle; human chorionic gonadotropin; progesterone; progesterone rise; ovulation
MeSH Terms: conditions — Infertility, Female | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pure Natural Cycle: * Transvaginal ultrasound (TVUS) on day 2/3 of cycle + hormones FSH, LH, E2, P4 (IVF1)
  * TVUS day 9-10 of cycle to identify dominant follicle.
  * Blood test for IVF1 every 24h until identification of the LH surge.
  * The LH surge will be diagnosed when the concentration rises by 180% above the latest serum value available in that patient and continued to rise thereafter (Fatemi et al, 2010).
  * Once the LH rise is detected, blood test for IVF1 to be performed after 2h, and then every 12h after LH rise for 2 days.
  * During luteal phase, IVF1 day 7 after LH rise and day 14 after LH rise.
- Modified Natural Cycle: * Transvaginal ultrasound (TVUS) on day 2/3 of cycle + hormones FSH, LH, E2, P4 (IVF1)
  * TVUS day 9-10 of cycle to identify dominant follicle.
  * Once the dominant follicle reaches 17mm or above, a bolus of 6500 rhCG (Ovitrelle, Merck-Serono) will be administered subcutaneously. IVF1 to be performed just before the rhCG-administration.
  * IVF1 2h after rhCG.
  * IVF1 every 12h for 2 days after rhCG.
  * During luteal phase, IVF1 day 7 after rhCG and day 14 after rhCG.
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — once the dominant follicle reaches 17mm or above, a bolus of 6500 rhCG (Ovitrelle, Merck-Serono) will be administered subcutaneously
  Other Names: Ovitrelle
  Groups: Modified Natural Cycle

SUMMARY:
Natural cycles are evaluated during fertility treatments for different therapeutic options, like insemination (IUI), time intercourse (TI) or frozen-thawed embryo transfers (FET). Two possible protocols can be used for natural cycles, with or without hCG trigger. Usually, studies including natural cycles consider both options as equivalent, not considering the possible bias that the exogenous hCG (human chorionic gonadotrophin) might have. In this prospective study, Investigators aim to evaluate the differences in the hormonal profile during the ovulation when it occurs spontaneously vs triggered with a bolus of hCG.

DETAILED DESCRIPTION:
For the pure natural cycle (PNC), ovulation will be detected by a combination of ultrasound monitoring the follicular growth and serial measurement of luteinizing hormone (LH), estradiol (E2) and progesterone (P4) levels, which is recognised to be the most accurate method of correctly identifying ovulation.

For the modified natural cycle (MNC), a bolus of rhCG 6500 IU subcutaneous (sc) will be administered when 1 dominant follicle reaches 17mm or above, after excluding previous LH surge. This is the first prospective study where the differences on the hormonal profile for ovulation will be studied.

HYPOTHESIS:

H0: The hormonal profile is not different between the PNC and the MNC H1: The hormonal profile is different between the PNC and MNC

Administration of hCG is a popular method for triggering ovulation since it may avoid the need to perform IUI or FET at weekends. However, it is an intervention compared with the detection of the spontaneous LH rise. Moreover, due to the presence of hCG receptors in the human endometrium, administration of hCG might interfere with endometrial receptivity. Previous publications evaluating pregnancy rates demonstrated that the use of hCG injection during the natural cycle reduces the pregnancy rates, in FET and IUI. It remains unclear what might be the mechanism to explain the lower pregnancy rates: a possible direct effect of hCG on the hCG receptors of the endometrium or a modification of the hormonal profile after the administration of the hCG, affecting the window of implantation (WOI).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women below 40 years
* Regular and Ovulatory cycles

Exclusion Criteria:

* Previous adnexal surgery
* Endometriosis
* PCOs
* Using hormonal contraception during the previous 2 months: OCP, progesterone IUD

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — healthy women with spontaneous ovulation
Study Population: healthy women with spontaneous ovulation
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Difference in hormone levels | 35 days
  Small sample data will be analyzed with the use of non-parametric test like Wilcoxon test to a paired a test of difference in hormones levels of the patients represented in both cycles (PNC and MNC) (dependent samples). This test will be preferred due to non-independent interval or ratio data in addition not to meet the normality or homogeneity of variances assumptions as paired t-test.
  Hormonal pattern over the days (measured for some days during cycle 1 and cycle 2) will be analyzed using trend analysis (line fit).

SECONDARY OUTCOMES:
Number of visits in luteal phase | 17 days
  Number of visits will be analyzed. The differences will be analyzed across PNC and MNC with CI. Fisher's exact test.
Luteal phase length | 17 days
  Luteal phase length will be analyzed. The differences will be analyzed across PNC and MNC with CI. Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: LAURA MELADO, PhD, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Licht P, Fluhr H, Neuwinger J, Wallwiener D, Wildt L. Is human chorionic gonadotropin directly involved in the regulation of human implantation? Mol Cell Endocrinol. 2007 Apr 15;269(1-2):85-92. doi: 10.1016/j.mce.2006.09.016. Epub 2007 Feb 14. PMID 17367920
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Background] Kyrou D, Kolibianakis EM, Fatemi HM, Grimbizis GF, Theodoridis TD, Camus M, Tournaye H, Tarlatzis BC, Devroey P. Spontaneous triggering of ovulation versus HCG administration in patients undergoing IUI: a prospective randomized study. Reprod Biomed Online. 2012 Sep;25(3):278-83. doi: 10.1016/j.rbmo.2012.05.005. Epub 2012 May 23. PMID 22796236
- [Background] Connelly LM. Pilot studies. Medsurg Nurs. 2008 Dec;17(6):411-2. No abstract available. PMID 19248407
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- See also: van Belle, G. (2002). Statistical rules of thumb. New York: John Wiley — http://vanbelle.org/presentations/CHSTalkNoPictures.pdf